CLINICAL TRIAL: NCT03612492
Title: The Effects of Lidocaine and Esmolol on Attenuation of Hemodynamic Response to Orotracheal Intubation: A Double-blind, Randomized, Clinical Trial
Brief Title: The Effects of Lidocaine and Esmolol on Attenuation of Hemodynamic Response to Orotracheal Intubation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, Preceptor of Medical Residency in Anesthesiology, Hospital de Base
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Esmolol vs Lidocaine on OTI
Record Dates: First submitted 2018-07-25; First posted 2018-08-02 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Hemodynamic Instability
Keywords: esmolol; lidocaine; intubation; hemodynamic response
MeSH Terms: interventions — esmolol; Adrenergic beta-Antagonists; Lidocaine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esmolol Group (Active Comparator): Patients will receive esmolol during induction of anesthesia
  Interventions: Drug: Esmolol; Drug: Lidocaine
- Lidocaine Group (Active Comparator): Patients will receive lidocaine during induction of anesthesia
  Interventions: Drug: Esmolol; Drug: Lidocaine

INTERVENTIONS:
Drug: Esmolol — Esmolol group (EG) will receive a bolus of esmolol 1.5mg / kg in 10 min following by continuous infusion at a rate of 0.1mg / kg / min.
  Other Names: Beta blocker
Drug: Lidocaine — Lidocaine (LG) group will received lidocaine bolus of 1.5mg / kg in 10 min following by continuous infusion at a rate of 1.5mg / kg / h.
  Other Names: Local anesthetic

SUMMARY:
The present study aims to compare the hemodynamic response during laryngoscopy and orotracheal intubation using continuous infusion of lidocaine and esmolol in patients undergoing general anesthesia.

DETAILED DESCRIPTION:
Esmolol is a selective beta-blocker of fast action that antagonizes beta-1 adrenergic receptors. Venous lidocaine is the agent most used to attenuate the hemodynamic response to laryngoscopy and intubation, in addition to cough reflex.

Objective: To compare the hemodynamic response during laryngoscopy and orotracheal intubation using continuous infusion of lidocaine and esmolol.

Methods: Randomized, double masked clinical trial aims to compare the effect of esmolol and lidocaine on orotracheal intubation. All patients will receive balanced general anesthesia. One group (EG) will receive bolus esmolol of 1.5mg / kg in 10 min following by continuous infusion at a rate of 0.1mg / kg / min. The lidocaine (LG) group will receive lidocaine bolus of 1.5mg / kg in 10 min following by continuous infusion at a rate of 1.5mg / kg / h.

Data on hemodynamic changes, reaction to laryngoscopy, conditions at intubation and adverse events will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years
* Physical State 1, 2 or 3 of the American Society of Anesthesiology (ASA)
* Electively or urgently scheduled for surgery requiring general anesthesia, with programming of orotracheal intubation via direct laryngoscopy at the Base Hospital of the Federal District.

Exclusion Criteria:

* Patients younger than 18 and over 70 years of age
* Patients with contraindications or history of hypersensitivity to the drugs involved in the study
* Patients with coronary ischemic disease
* Patients with atrioventricular block at any grade
* Patients with diagnosed cardiac arrhythmias
* Patients with heart failure
* Patients who are beta-blockers or calcium channel blockers
* Patients with renal insufficiency of any kind
* Patients with difficulty predicting orotracheal intubation
* Patients with BMI ≥ 35 kg / m²
* Patients who underwent neuroaxis block before anesthetic induction
* Patients who refuse to participate in the study after submitting the informed consent form
* Patients requiring two or more attempts of laryngoscopy for positioning of the orotracheal tube
* Patients with asthma
* Any other condition that, in the opinion of the researcher, may pose a risk to the patient or interfere with the objectives of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with tachycardia after intubation | 12 minutes
  Analysis of the incidence of tachycardia after intubation

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 12 minutes
  Hemodynamic stability analysis through the incidence of tachycardia, hypertension, bradycardia, hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Singh S, Laing EF, Owiredu WK, Singh A. Comparison of esmolol and lidocaine for attenuation of cardiovascular stress response to laryngoscopy and endotracheal intubation in a Ghanaian population. Anesth Essays Res. 2013 Jan-Apr;7(1):83-8. doi: 10.4103/0259-1162.114008. PMID 25885726
- [Background] Mendonca FT, de Queiroz LM, Guimaraes CC, Xavier AC. Effects of lidocaine and magnesium sulfate in attenuating hemodynamic response to tracheal intubation: single-center, prospective, double-blind, randomized study. Braz J Anesthesiol. 2017 Jan-Feb;67(1):50-56. doi: 10.1016/j.bjane.2015.08.004. Epub 2016 Nov 22. PMID 28017170